CLINICAL TRIAL: NCT00448825
Title: Novel Pharmacotherapy for Dual Dependence
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bankole Johnson (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Bankole Johnson, Chair of Psychiatry and Neurobehavioral Sciences, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11620; R01DA019804 (NIH); DPMCDA (Other: NIDA)
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Alcohol Dependence; Cocaine Dependence
Keywords: alcohol dependence; alcoholism; cocaine addiction; cocaine dependence
MeSH Terms: conditions — Alcoholism; Cocaine-Related Disorders | interventions — Topiramate; Cognitive Behavioral Therapy; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Experimental): Topiramate + Cognitive Behavioral Therapy
  Interventions: Drug: Topiramate + Cognitive Behavioral Therapy
- Placebo (Placebo Comparator): Placebo + Cognitive Behavioral Therapy
  Interventions: Drug: Placebo + Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Topiramate + Cognitive Behavioral Therapy — Topiramate up to 300 mg per day
  Other Names: Topamax
  Arms: Topiramate
Drug: Placebo + Cognitive Behavioral Therapy — Placebo twice a day
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of Topiramate and Cognitive Behavioral Therapy for the treatment of alcohol and cocaine dependence.

DETAILED DESCRIPTION:
Our objective is to understand the basic mechanisms that underpin substance dependence, and to develop efficacious treatments for individuals with comorbid cocaine and alcohol dependence.

Participants in this study will be randomly assigned to receive either 300 mg per day of topiramate or placebo. In addition, participants will receive weekly cognitive behavioral therapy for 12 weeks.Follow-up visits will occur at 2 weeks and 1,2,, and 3 months following completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be men and women between the ages of 18 years and older.
* Must meet at least three of the seven DSM IV diagnostic criteria for alcohol and cocaine dependence.
* Express a desire for treatment.
* Literacy in English and ability to read, understand, and complete the ratings scales and questionnaires accurately, follow instructions, and make use of the behavioral treatments are required.
* Prospective subjects must report cocaine use of at least once per month and alcohol consumption of ≥21 drinks/week and ≥14 drinks/week for men and women respectively, during the past 30 days
* At least one positive urine drug screen for cocaine at screen or baseline prior to randomization.

Exclusion Criteria:

Please contact site for additional information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2007-03; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
The topiramate group will be superior to the placebo group on the following outcome measures:increasing the weekly mean proportion of cocaine-free days, decreasing self-reported drinking, and decreasing craving for cocaine and alcohol. | According to Preston Rules from weeks 6 to 12.
  Alcohol - assessed by self-report of use (TLFB,DD,DDD,PDA, PHDD), biochemical markers (GGT, CDT), OCDS
  Cocaine - assessed by self-report of use (CTFB, substance use inventory, QFI),urine assay for benzoylecgonine, and CCQ-NOW

SECONDARY OUTCOMES:
a. Cocaine free weeks; b. Topiramate, compared with placebo, will be associated with an improvement in psychosocial functioning as exemplified by improved general well-being, social functioning, and quality of life. | According to Preston Rules from weeks 1 to 12
  1. Cocaine free weeks is assessed by a combination of self-report of use and urine assays;
  2. Assessed by increased scores in the following assessments: CGI, BSI, Q-LES-Q, DrInC, SFQ, medication compliance, CIWA-Ar, POMS, BIS

CONTACTS AND LOCATIONS:
Overall Officials: Bankole Johnson, DSc, MD, PhD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - University of Virginia Center for Addiction Research and Education, Charlottesville, Virginia
  - University of Virginia Center for Addiction Research and Education, Richmond, Virginia